CLINICAL TRIAL: NCT06286371
Title: Pelvic Neuro-Angiogenesis Density in the Presence of Deep Endometriosis and Relationship Between Pelvic Pain Scores
Brief Title: Pelvic Neuro-Angiogenesis in Deep Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, GÜRKAN UNCU,PROF. MD, Prof., Uludag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-13/37
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis-related Pain; Endometriosis; Deep Endometriosis; Endometriosis; Peritoneum
Keywords: Endometriosis; Deep Endometriosis; Pelvic Pain; Neurogenesis; Endometriotic Nodule; Laparoscopy; Endometriosis Surgery
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): This study has only one group, the group includes patients with laparoscopic endometriosis surgery (douglasectomy).
  Interventions: Procedure: Laparoscopic Endometriosis Surgery

INTERVENTIONS:
Procedure: Laparoscopic Endometriosis Surgery — Laparoscopic Excision of Deep Endometriotic Nodule related to pelvic pain

SUMMARY:
Endometriosis is observed in one out of every ten women in society, causing endometrial cells to be found outside their normal location in the body and proliferate in other locations, leading to fibrosis in the tissue due to the secretion of various factors from the cells. Additionally, the substances secreted by the cells can cause various other changes in the tissue besides fibrosis. Increased neurogenesis and neovascularization are among the primary changes, which occur as a result of the secretion of substances from the cells. Increased neovascularization, neurogenesis, and fibrosis in the tissue lead to the formation of nodular structures in the pelvic region, resulting in pain development in women.

Nodular formations in the pelvic region due to endometriosis are especially observed in the rectovaginal space. Despite being small in size, they can induce increased neovascularization and neurogenesis even in healthy peritoneal tissue due to the microenvironment they create, leading to different clinical symptoms clinically. However, it is not known how far these changes occur around the endometriotic nodule in the presence of endometriosis.

In this project, in patients operated on due to endometriosis, the density of nerve and vascular structures in the surgical margins of the peritoneal tissue excised along with the nodule, and the synthesis and release of chemical mediators causing pain (e.g., Bradykinin, Substance-P) are evaluated. The aim is to determine the minimum surgical margin where excision should be applied in surgery and to demonstrate any endometriotic changes that may exist in the tissues, even though they may appear macroscopically healthy.

DETAILED DESCRIPTION:
This study aims to investigate the relationship between the neurovascular density and the amount of pain mediators present in the excised endometriotic nodule and peritoneal surface during laparoscopic douglasectomy surgery routinely performed in cases of endometriosis unresponsive to medical treatment, and their correlation with pain scores. Together with the findings obtained, the goal is to determine the excision boundaries and surgical safe margins in endometriosis surgery.

Since endometriosis primarily affects the pelvic region, women often encounter various types of chronic pelvic pain, dyspareunia, dysmenorrhea, and dyschezia in daily life depending on the size and location of the nodule, which do not pass frequently. These pains often do not respond to analgesic drugs, and patients experience severe pain attacks. As it is a disease dependent on estrogen in treatment, treatments containing anti-estrogenic and progesterone are primarily applied to suppress the development of endometriosis, while the surgical removal of endometriotic nodules in cases unresponsive to medical treatment provides benefit in terms of pain palliation. In this context, although surgery ideally performed as laparoscopic surgery, peritoneal nodules in the pelvic region are excised together, a procedure called douglasectomy. In many animal experiments, endometriosis nodules have been histopathologically examined, and it has been shown that there is a rich structure in terms of nerve fibers, vascular structure, and pain mediators within the nodule. However, this surgery is a highly specific surgical method and is performed by experienced centers and surgeons. Consequently, the number of patients undergoing ideal surgery is limited. In this limited population, the vascular and neurogenic structure in the peritoneum and nodule surgically removed after douglasectomy, as well as the amount of pain mediators synthesis, remains an unexplored virgin subject. Although increased nerve density within the nodule has been shown in limited studies, the clinical relationship of this density, and its effects on pain scores, has not been investigated in any study on the pathology material removed after douglasectomy operation.

Through the data obtained from this research, the investigators will conclude the histological boundaries of neuro-angiogenic changes occurring in endometriosis disease, the extent of involvement in the pelvic peritoneum, and thus the minimum amount of tissue to be excised during surgery. This result will shed light on a topic that has not been studied in the literature so far and will be a milestone in terms of excision boundaries and surgical safe margins in endometriosis surgery.

This clinical study, approved by the Bursa Uludağ University Faculty of Medicine Clinical Research Ethics Committee with decision number 2023-13/37 on 13.06.2023, will be conducted in the Department of Obstetrics and Gynecology at Bursa Uludağ University Faculty of Medicine. Women of reproductive age who apply to the endometriosis clinic, cannot respond to medical treatment, and are planned for surgery will be included in the study. An average of approximately 150 endometriosis surgeries are performed in our clinic annually. The number of patients to be included in the study was calculated as at least 15 in the power analysis conducted, and the patient recruitment for the study will be completed in a short time in our center, where approximately 150 endometriosis surgeries are performed annually. All demographic data of the patients, preoperative laboratory, and clinical findings will be recorded through files. From the patients who agree to participate in the study, peritoneal tissue samples of 1 cm in size (Figure-1) taken from the pathology specimen removed after the routine surgical procedure will be histopathologically examined, and nerve fibers and vascular structures per square millimeter will be counted after appropriate staining (hematoxylin & eosin and toluidine blue). In addition, tissue samples preserved under appropriate conditions will be examined for pain mediators (bradykinin, substance P, nerve growth factor, PGP9.5) using the ELISA (Enzyme-Linked ImmunoSorbent Assay) method with kits to be obtained. An average of 10 peritoneal tissue samples will be taken from each patient, and a total of 150 samples will be examined. Each sample will be analyzed twice using the ELISA method, and at least 4 sets of 96 kits will be required for the examination of mediators in 150 separate tissue samples. Results will be analyzed following the commercial ELISA kit protocol. Through the obtained data, the correlation between preoperative pain scores (VAS score - visual pain score) and the neurovascular density within the nodule will be evaluated, and the effects of laparoscopic surgery with nodule excision on pain will be histopathologically demonstrated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion of deep endometriosis (Physical Examination and MRI)
* Patients with ineffective response to medical therapy
* Patients who undergo laparoscopic conservative endometriosis surgery (douglasectomy)

Exclusion Criteria:

* Patients with malignity suspicion
* Patients with extensive surgery (hysterectomy, ovariectomy)
* Patients with previous endometriosis or another pelvic surgery
* Patients with oocyte pick up procedure history
* Patients with pelvic inflammatory disease history

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Density of Neuro-Angiogenesis | 6 months
  Density of nerve fibers and capillaries in each 1 cm peritoneal leaf which excised during laparoscopic endometriosis surgery
Density of Pain Mediators in Pelvic Peritoneum | 6 months
  Density of Substance-P, Bradykinin, Nerve Growth Factor and PGP 9.5 in each peritoneal leaf which excised during surgery

SECONDARY OUTCOMES:
Relationship between Neuro-Angiogenesis Density and Pelvic Pain Scores | 6 months
  Patients will be surveyed before and after (0., 3., 6. months) surgery about the visual analogue scores for pelvic pain, and the scores will be analyzed to determine if there is any correlated factor (nerve density, capillary denstiy or pain mediators) with pelvic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Gurkan Uncu, Prof., Study Chair — Uludag University
Locations (1):
- Uludag University Faculty Hospital, Bursa, Gorukle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No